CLINICAL TRIAL: NCT05757115
Title: Evaluation and Development of Playing Skills for Parents With Children With Special Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Zeynep Çorakcı Yazıcıoğlu, Principal Investigator, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CORAKCİ-002
Record Dates: First submitted 2023-02-06; First posted 2023-03-07 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Play and Playthings
Keywords: Neurodevelopmental Disorders, Autism Spectrum Disorders, Parents, Mentoring, Play and Playthings
MeSH Terms: conditions — Neurodevelopmental Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Parents with children with special needs who want to participate in the study will be determined. The assessments will be applied to parents before and after play training. These trainings aim to develop the skills of playing games with their children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): It is the group to which individualized training will be applied to develop play skills.
  Interventions: Behavioral: Play Skills Training

INTERVENTIONS:
Behavioral: Play Skills Training — Each parent will be provided with "play skills training" that will support them to spend effective and meaningful time with their child. While planning the educational contents, an Occupational Therapy Model suitable for the parent and the child will be used. The process will be followed by giving unique recommendations to each parent. Recommendations given based on feedback will be revised.

SUMMARY:
Children with special needs; experiences physical, behavioral, social, cognitive and emotional limitations. These limitations affect the child's play skills. They need to be supported and encouraged by their parents to enable them to participate in the game. Parental playing skills creativity, self-efficacy and active participation are important factors in this regard.

In current studies, parents with special needs children; It is supported that there is a relationship between play, acting and parental self-efficacy. In this study, it was aimed to improve the skills of parents with special needs children to play games with their children multidimensionally and to develop these skills with individual-specific techniques.

Detailed assessments will be carried out in order to determine the functional, cognitive and psychosocial skills of the parents.

After the evaluation phase is completed, the scores of each parent will be analyzed and interpreted according to Occupational Therapy Models. Playing training will be given individually according to parameters such as strong and weak features, strong sensory system, personality traits, predisposition and defensive approaches.

ELIGIBILITY:
Inclusion Criteria:

* Being a mother of a special needs child
* The age of her child is 2-6 years
* Being able to speak Turkish
* Volunteer to participate in the study

Exclusion Criteria:

* Have training in play therapy
* Having a psychiatric or neurological disease that significantly affects cognitive status

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mothers of children with special needs will be included
Enrollment: 17 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Adult Playfulness Trait Scale | 2 mounths
  The scale consists of 19 items. Each item falls under one of the three subscales: funseeking motivation, uninhibitedness and spontaneity. All items were randomly ordered and used seven-point likert scales with all points labeled (1= "strongly disagree", 7= "strongly agree").

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It is aimed to share all the collected individual participant data in a scientific publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 6 months after publication
Access Criteria: Can be shared with researchers working with similar keywords